CLINICAL TRIAL: NCT01477216
Title: The Glycemic and Insulinemic Responses of the Finnish Foods: Measurement and Modification
Brief Title: Determination of Glycemic and Insulinemic Indices
Acronym: ELSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: TUSU 182-5
Record Dates: First submitted 2011-10-04; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Glucose Metabolism
Keywords: Glycemic index; Glycemic responses; Insulin responses; Insulinemic index; Carbohydrates; Methodology; Glucose metabolism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (9):
- Measuring method (Experimental): To compare glycemic responses and GI values from capillary and venous blood and to compare glucose solution with white bread as the reference food and to study the effect of the number of reference tests on GI values.
  Interventions: Other: ELSA 1-9
- Mixed meals (Experimental): To examine the glycaemic and insulinaemic responses of a mashed potato-based meal when a high fat food (rapeseed oil) or a high protein food (chicken breast) or fat, protein and salad together were added to the meal. Furthermore, we studied how the predicted and measured GI values of the mixed meal differed from each other.
  Interventions: Other: ELSA 1-9
- Coffee (Experimental): To examine the effects of two different coffee portions with glucose and caffeine-containing soft drinks on postprandial glucose and insulin responses. Further objectives were to study how coffee and different accompaniments affect glucose and insulin responses.
  Interventions: Other: ELSA 1-9
- Snacks (Experimental): To measure GI and II values for Finnish snack foods
  Interventions: Other: ELSA 1-9
- Berries (Experimental): To study the effects of berries on glycemic and insulinemic responses
  Interventions: Other: ELSA 1-9
- GIs of low-carbs (Experimental): To measure glycemic and insulinemic responses to low-carbohydrates foods
  Interventions: Other: ELSA 1-9
- Glucose metabolism and BMI (Experimental): To examine the effects of overweight and glucose tolerance on the glucose, insulin and lipid responses to an HGI meal and an LGI meal. Furthermore, the second aim was to study the effect of BMI and glucose tolerance on the GI measured.
  Interventions: Other: ELSA 1-9
- Insulin measurement (Experimental): To compare how methodological choices affect measured insulin values
  Interventions: Other: ELSA 1-9
- Alcohol (Experimental): To investigate the effect of alcohol on postprandial glucose and insulin responses, and to determine glycemic and insulinemic indices values for beer and non-alcoholic beer.
  Interventions: Other: ELSA 1-9

INTERVENTIONS:
Other: ELSA 1-9 — Measuring GI and II values for Finnish foods

SUMMARY:
The aim of this study to investigate methodological aspects that may affect glycemic index (GI) and insulinemic (II) values. In addition, we will measure GI and II values for typical Finnish carbohydrate-rich foods and provide a database of GIs for Finnish foods.

The specific aims of this study are:

* to compare glycemic responses and GIs analyzed from capillary and venous blood to compare glucose against white bread as the reference food, and to study the effect of number of reference tests on GI values. For each setting of the tested parameters, we determined the glycemic indices of rye bread, oatmeal porridge and instant mashed potato
* to examine the glycaemic and insulinaemic responses of a mashed potato-based meal when a high fat food (rapeseed oil) or a high protein food (chicken breast) or fat, protein and salad together were added to the meal. Furthermore, we studied how the predicted and measured GI values of the mixed meal differed from each other.
* to examine the effects of two different coffee portions with glucose and caffeine-containing soft drinks on postprandial glucose and insulin responses. Further objectives were to study how coffee and different accompaniments affect glucose and insulin responses.
* to measure GI values for typical Finnish foods
* to study the effects of berries on glycemic and insulinemic responses
* to examine the effects of overweight and glucose tolerance on the glucose, insulin and lipid responses to an HGI meal and an LGI meal.Furthermore, the second aim was to study the effect of BMI and glucose tolerance on the GI measured.
* to compare methodological choices in insulin measurement
* to investigate the effect of alcohol on postprandial glucose and insulin responses, and to determine glycemic and insulinemic indices values for beer and non-alcoholic beer

ELIGIBILITY:
Inclusion Criteria:

* For Studies 1-9 a total of 12 to 24 volunteers per study with a normal glucose tolerance based upon a 2 h 75g oral glucose tolerance test (OGTT).
* For Study 7 a total of 24 volunteers with impaired glucose tolerance based on an OGTT.
* For Studies 1-6 and 8-9 with an age of 20 to 60 and with a BMI of 18 to 30 kg/m2.
* For Study 7 an age of 62 to 72 and with a BMI of 20 to 35 kg/m2.

Exclusion Criteria:

* First-degree family history of diabetes
* An active gastrointestinal or metabolic disease
* For Studies 1-6 and 8-9 chronic medication (oral contraceptives were allowed)
* For Study 7 regular medication that would have affect glucose and lipid metabolism
* Smoking
* Pregnancy
* Breastfeeding
* History of polycystic ovary syndrome
* History of gestational diabetes

Ages: 20 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2003-01; Primary Completion 2008-12 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Glucose | 2 to 5 hours
  Area under the plasma concentration versus time curve (AUC) of food
Insulin | 2 to 5 hours
  Area under the plasma concentration versus time curve (AUC) of food
Free fatty acids | 2 to 5 hours
  Area under the plasma concentration versus time curve (AUC) of food
Triglyserides | 2 to 5 hours
  Area under the plasma concentration versus time curve (AUC) of food

SECONDARY OUTCOMES:
IGF1 | 2 to 5 hours
  Area under the plasma concentration versus time curve (AUC) of food
Satiety | 2 to 5 hours
  Satiety scores on the satiety scale
IGF-BP1 | 2 to 5 hours
  Area under the plasma concentration versus time curve (AUC) of food

CONTACTS AND LOCATIONS:
Overall Officials: Liisa M Valsta, DSc, Study Director — National Institute for Health and Welfare, Helsinki, Finland; Katja A Hätönen, Principal Investigator — National Institute for Health and Welfare, Helsinki, Finland

REFERENCES:
- [Derived] Hatonen KA, Virtamo J, Eriksson JG, Perala MM, Sinkko HK, Leiviska J, Valsta LM. Modifying effects of alcohol on the postprandial glucose and insulin responses in healthy subjects. Am J Clin Nutr. 2012 Jul;96(1):44-9. doi: 10.3945/ajcn.111.031682. Epub 2012 May 30. PMID 22648716